CLINICAL TRIAL: NCT01197274
Title: Comparison of Simple Blood Lancet(Vitrex®)With DuoTip as Devices for Skin Prick Test Among Mite-sensitized Subjects
Brief Title: Comparison of Simple Blood Lancet(Vitrex®)With DuoTip as Skin Prick Test Devices Among Mite-sensitized Subjects
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Professor Pakit Vichyanond, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University
Other Study IDs: 186/2553(EC4)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-06

CONDITIONS: Skin Prick Test
Keywords: allergy; skin prick test; mite sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mite-sensitized person
  Interventions: Device: Simple blood lancet

INTERVENTIONS:
Device: Simple blood lancet — Skin prick testing with blood lancet and DuoTip is performed on the back of mite-sensitized person. Allergen(Der p)is placed in 1st and 2nd row whereas histamine is placed in 3rd row. Allergen and normal saline are placed alternately in 4th row. Block randomization were allocated subjects into 2 groups; Group1:blood lancet is performed in 1st row and DuoTip in 2nd row. Group2:DuoTip is performed in 1st row and blood lancet in 2nd row. Blood lancet is applied in 3rd and 4th row in all subjects. A technician performed device applications and another technician who is blinded to device performed all readings. Pain was assessed on a scale from 0 to 10 with 0 being no pain and 10 being the worst imaginable pain
  Other Names: Vitrex®

SUMMARY:
The purpose of this study is to compare the results skin prick tests using simple blood lancet (Vitrex®) with DuoTips among mite-sensitized subjects.

DETAILED DESCRIPTION:
We intend to compare results of skin prick tests by using simple blood lancet(Vitrex®) and DuoTips in terms of wheal size, variability, transfer of allergen and pain level, among mite-sensitive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Who have positive skin prick testing to Der p 10,000 AU/ml (wheal size 3 mm at least)
* Age 12-60 yrs
* Written informed consent was obtained from all subjects and their parents

Exclusion Criteria:

* Who have positive skin prick testing to Der p 10,000 AU/ml above 15 mm.
* Who have dermographism
* Who have severe disease eg. severe respiratory disease or severe cardiovascular disease
* Who have severe eczema
* Who receive antihistamine, topical steroid within 7 days or ketotifen within 14 days or systemic steroid within 1 month
* Pregnant women

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals who have positive skin prick testing to Der p 10,000 AU/ml (wheal size 3 mm at least)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Wheal and flare reaction to Der p results of skin prick test by simple blood lancet (Vitrex®) | 15 minutes
  To determine
  1. Wheal and flare diameter to Der p performed by blood lancet(Vitrex®)compared with DuoTip in mite-sensitized person
  2. Intradevice variability or coefficients of variation of blood lancet compared wtih DuoTip

SECONDARY OUTCOMES:
Determine transfer of allergen by simple blood lancet and Duotips. | 15 minutes
  To determine
  1. Transfer of allergen(Der p)performed by simple blood lancet(Vitrex®)
  2. Pain assessment by using visual analog scale
  3. Wheal and flare diameter to histamine performed by simple blood lancet(Vitrex®)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Pakit Vichyanond, MD, Study Director — Siriraj Hospital
Locations (1):
- Department of Pediatrics, Siriraj hospital, Mahidol University, Bangkok, Thailand